CLINICAL TRIAL: NCT03823404
Title: GAIN Trial: A Randomized, Double-Blind, Placebo-Controlled Study of COR388 in Subjects With Alzheimer's Disease
Brief Title: GAIN Trial: Phase 2/3 Study of COR388 in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cortexyme Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR388-010
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — COR388

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- COR388 80 mg twice daily (BID) (Experimental): COR388 hydrochloric acid (HCl), 80 mg orally administered capsule, BID (twice daily) with water approximately 12 hours apart and no less than 6 hours apart
  Interventions: Drug: COR388 capsule
- COR388 40 mg BID (Experimental): COR388 HCl, 40 mg orally administered capsule, BID with water approximately 12 hours apart and no less than 6 hours apart
  Interventions: Drug: COR388 capsule
- Placebo BID (Placebo Comparator): Placebo orally administered capsule, BID with water approximately 12 hours apart and no less than 6 hours apart
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: COR388 capsule — BID (twice daily)
  Other Names: atuzaginstat
  Arms: COR388 40 mg BID; COR388 80 mg twice daily (BID)
Drug: Placebo capsule — BID
  Other Names: atuzaginstat
  Arms: Placebo BID

SUMMARY:
This is a randomized, double-blind, placebo-controlled study that assessed the efficacy, safety, and tolerability of 2 dose levels of COR388 in subjects with a clinical diagnosis of mild to moderate Alzheimer's disease (AD) dementia.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study that assessed the efficacy, safety, and tolerability of 2 dose levels of COR388 oral capsules in subjects with probable Alzheimer's disease (AD) dementia according to the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria. The subject did not have other conditions or brain imaging abnormalities that could explain the symptoms of dementia. All subjects were encouraged to have lumbar punctures (LPs) (during screening, week 24 and week 48) in the absence of medical conditions that could increase the risk of the procedure in the opinion of the Investigator. Cerebrospinal fluid (CSF), saliva, and blood were analyzed for measurements of biomarkers of AD and neuroinflammation, and for the presence of bacterial deoxyribonucleic acid (DNA) of Porphyromonas gingivalis (P. gingivalis). A subset of sites monitored subjects for clinical evidence of periodontitis at baseline, 24 and 48 weeks.

The study consisted of 3 phases: a screening phase of up to 6 weeks, a treatment phase of up to 48 weeks, and a safety follow-up phase of 6 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has probable AD dementia according to the NIA-AA criteria.
* Subject has an Mini-Mental State Examination (MMSE) score 12 and 24 inclusive at both screening and Visit 2 and a ≤3-point difference between these visits.
* Subject has brain MRI scan consistent with the diagnosis of AD performed during the screening period. Computed Tomography scan can be used only if the subject has an absolute contraindication for MRI.
* Subject has a Modified Hachinski score ≤4 at screening.
* Subjects with background symptomatic therapy with acetylcholine esterase inhibitors, and/or memantine, are allowed as long as the dose has been stable for 90 days prior to screening and no changes are planned during the study.
* Subject has a primary caregiver willing to accept responsibility for supervising the treatment (e.g., administering study drug) and assessing the condition of the subject throughout the study in accordance with all protocol requirements.
* Subject has body mass index <38 kg/m2 at Screening

Key Exclusion Criteria:

* Subject has imaging consistent with a dementia diagnosis other than AD.
* Subject has had an increase or restoration of cognition based on medical history.
* Subject with history or current evidence of major psychiatric illness such as schizophrenia, bipolar disorder, or major depressive disorder that may interfere with the patient's ability to perform the study and all assessments. Note: Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. The use of anti-depressants or the use of anti epileptic medication for non seizure-related treatment is allowed if the dose has remained stable for at least 60 days prior to enrollment.
* Subject has any of the following laboratory findings at screening:

  1. Alanine aminotransferase >3 x upper limit of normal (ULN), aspartate aminotransferase >3 x ULN, or history of clinically significant liver disease in the Investigator's judgment.
  2. Hemoglobin ≤10 g/dl.
  3. Creatinine clearance (CL) of <45 ml/min.
  4. Poorly controlled diabetes as defined by hemoglobin A1C (HbA1C) >8.
  5. Positive blood screen for Human Immunodeficiency Virus (HIV 1 and 2), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus antibodies (HCV-Ab) at Screening.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female.
Enrollment: 643 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Smith, MD, Study Director — Quince Therapeutics Inc
Locations (93):
- United States (58):
  - Xenoscience, Inc., Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health, Sun City, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Alliance Research, Long Beach, California
  - Standford University, Palo Alto, California
  - CITRIALS, Riverside, California
  - CITRIALS, Santa Ana, California
  - Syrentis Clinical Research, Santa Ana, California
  - Southern California Research LLC, Simi Valley, California
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Qtrials, Inc., Miami, Florida
  - Future Care Solutions, LLC, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Bioclinica Research, Orlando, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Brain Matters Research at the Kane Center, Stuart, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Columus Memory Center, Columbus, Georgia
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Alexian Brothers Neurosciences Research, Elk Grove Village, Illinois
  - Ascension Via Christi Research, Wichita, Kansas
  - Activmed Practices and Research, Methuen, Massachusetts
  - The Boston Center for Memory, Newton, Massachusetts
  - Anil Nair MD, Alzheimer's Disease Center, Quincy, Massachusetts
  - Memory Center, Hattiesburg, Mississippi
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Princeton Medical Institute, Princeton, New Jersey
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - Neurology Specialists of Monmouth County, West Long Branch, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Disease Research & Neurology Center of Neurological Associates of Albany, Albany, New York
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Spri Clinicaltrials, Llc, Brooklyn, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - ANI Neurology, PLLC dba Alzheimer's Memory Center, Charlotte, North Carolina
  - Insight Clinical Trials, LLC, Beachwood, Ohio
  - Neurology Diagnostics Inc., Dayton, Ohio
  - Memory Health Center at Summit Research Network, Portland, Oregon
  - Northeastern Pennsylvania Memory and Alzheimer's Center, Plains, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Research Center, Dallas, Texas
  - Neurology Consultants of Dallas, Dallas, Texas
  - Houston Methodist Department of Neurology, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - University of Virginia Adult Neurology, Charlottesville, Virginia
  - Recognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - UW Alzheimer's Disease Research Center, Seattle, Washington
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- France (6):
  - Hôpital de Brabois, Toulouse, Cedex
  - Centre de Ressources Biologiques, Lille
  - University Hospital La Timone, Department of Neurology and Neuropsychology, Marseille
  - Service de Gériatrie, Nice
  - Hôpitaux Universitaires de Strasbourg, Centre d'Investigation Clinique, Hôpital Hautepierre, Strasbourg
  - CHRU de Nancy Hôpital de Brabois Service de Gériatrie, Vandœuvre-lès-Nancy
- Netherlands (5):
  - Brain Research Center Den Bosch B.V., 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - PreCare Trial & Recruitment, Beek
  - Isala Zwolle - Interne geneeskunde Centrum voor ouderengeneeskunde, Zwolle
  - Brain Research Center Zwolle, Zwolle
- Poland (7):
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - Krakowska Akademia Neurologii, Krakow
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie
  - Euromedis Sp. z o.o., Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - NZOZ Wrocławskie Centrum Alzheimerowskie, Wroclaw
- Spain (8):
  - Policlinica Gipuzkoa, San Sebastián, Gipuzkoa
  - Hospital General de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Fundacio Ace, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Marqués de Valdecilla, Santander
- United Kingdom (9):
  - Cognition Health Birmingham (private), Edgbaston, Birmingham
  - St Pancras Clinical Research (private), Barbican, London
  - Cognition Health Plymouth, Plymouth, Science Park
  - Memory Assessment and Research Centre, Moorgreen Hospital, Southampton, UK
  - RICE - The Research Institute for the Care of Older People, Bath
  - Glasgow Memory Clinic, Glasgow
  - Cognition Health Ltd. (private) Guildford, Guildford
  - Cognition Health Ltd. (private) London, London
  - Kingshill Research Centre Swindon, Swindon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 89 centers worldwide screened subjects and included 57 centers in the United States, 9 centers in the United Kingdom, 8 centers in Spain, 7 centers in Poland, 5 centers in France, and 3 centers in the Netherlands.
Pre-assignment Details: Randomized subjects were stratified by baseline Mini-Mental State Examination (MMSE) score (MMSE ≥12 and ≤18, and MMSE ≥19 and ≤24) and Apolipoprotein E genotype (ApoE4 positive either homozygous or heterozygous vs. all others) to assure balanced distribution of mild and moderate Alzheimer's disease and a balanced distribution of ApoE4 subjects, across treatment arms.
Groups:
- COR388 80 mg BID (Twice Daily); COR388 40 mg BID (Twice Daily): COR388 capsule: BID
- Placebo BID (Twice Daily): Placebo capsule: BID
Period: Overall Study
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Started | 214 | 212 | 217
Completed | 129 | 127 | 163
Not Completed | 85 | 85 | 54
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Adverse Event | 35 | 38 | 8
Not completed — Withdrawal by Subject | 38 | 40 | 35
Not completed — Death | 4 | 0 | 0
Not completed — Other: Various reasons provided | 5 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily) | Total
Number analyzed (Participants) | 214 | 212 | 217 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] — Age = age at consent
  years | 69.3 (6.9) | 68.6 (6.9) | 69.5 (6.9) | 69.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 123 | 125 | 365
  Male | 97 | 89 | 92 | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 18 | 25 | 78
  Not Hispanic or Latino | 174 | 188 | 187 | 549
  Unknown or Not Reported | 5 | 6 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 13 | 12 | 17 | 42
  White | 194 | 188 | 192 | 574
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 6 | 17
Region of Enrollment [Number; unit: participants]
  Netherlands | 10 | 13 | 8 | 31
  United States | 152 | 143 | 152 | 447
  Poland | 11 | 22 | 21 | 54
  United Kingdom | 24 | 12 | 13 | 49
  France | 10 | 8 | 10 | 28
  Spain | 7 | 14 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11)
Description: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11) - Total Score The cognitive subscale of the ADAS (ADAS Cog11) was used as a primary efficacy measure and consists of 11 items assessing areas of function most typically impaired in Alzheimer's disease (AD): orientation, verbal memory, language, and praxis. he scale ranges from 0 to 70, with higher scores indicating greater disease severity.
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 211 | 217
score on a scale
  Baseline | 23.7 (8.8) | 23.4 (8.6) | 23.6 (9.3)
  Average of Weeks 40/48: number analyzed (Participants) | 146 | 148 | 187
  Average of Weeks 40/48 | 26.6 (12.0) | 27.9 (11.8) | 28.4 (12.2)
Statistical Analysis 1: Comparison: COR388 80 mg BID (Twice Daily) vs COR388 40 mg BID (Twice Daily) vs Placebo BID (Twice Daily); Test type: Superiority; p < 0.0455, mixed-effects model for repeated measure — The interim analysis was conducted at significance level of 0.05 and the significance level was adjusted for final analysis

2. Primary Outcome: Alzheimer's Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL)
Description: The Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Inventory Score is a 23-item inventory.
  The ADCS-ADL measures both basic and instrumental activities of daily living The total ADCS-ADL score ranges from 0 to 78, with lower scores indicating greater disease severity.
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 211 | 217
score on a scale
  Baseline | 59.9 (11.2) | 60.1 (11.3) | 60.4 (11.3)
  Average of Weeks 40/48: number analyzed (Participants) | 149 | 150 | 188
  Average of Weeks 40/48 | 55.4 (13.9) | 54.4 (13.7) | 55.5 (14.1)
Statistical Analysis 1: Comparison: COR388 80 mg BID (Twice Daily) vs COR388 40 mg BID (Twice Daily) vs Placebo BID (Twice Daily); Test type: Superiority; p < 0455, Mixed Models Analysis

3. Secondary Outcome: Clinical Dementia Rating-Sum of Boxes (CDR-SB)
Description: Clinical Dementia Rating-Sum of Boxes (CDR-SB) - Sum of Boxes CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care.
  Severity score assigned for each of 6 domains; total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity.
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 211 | 217
score on a scale
  Baseline | 5.7 (2.6) | 6.0 (2.7) | 5.9 (2.8)
  Average of Weeks 40/48: number analyzed (Participants) | 149 | 150 | 188
  Average of Weeks 40/48 | 7.2 (3.6) | 7.2 (3.4) | 7.4 (3.5)

4. Secondary Outcome: Mini-Mental State Examination (MMSE)
Description: Change in Mini-Mental State Examination (MMSE) - Total Score Minimum Score - 0 Maximum Score - 30 Higher score means better outcome
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 212 | 217
score on a scale
  Baseline | 18.3 (3.3) | 18.4 (3.2) | 18.2 (3.3)
  Average of Week 40/48: number analyzed (Participants) | 146 | 149 | 186
  Average of Week 40/48 | 16.9 (5.7) | 16.4 (5.7) | 16.2 (5.9)

5. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: Neuropsychiatric Inventory (NPI) - Total Score NPI assesses psychopathology in participants with dementia and other neurologic disorders.
  Total score ranges from 12 to 144; higher scores indicate greater disease severity.
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 213 | 212 | 216
score on a scale
  Baseline | 6.7 (8.7) | 8.2 (11.2) | 8.1 (10.6)
  Average of Weeks 40/48: number analyzed (Participants) | 143 | 142 | 182
  Average of Weeks 40/48 | 10.7 (13.7) | 9.2 (12.1) | 10.4 (13.9)

6. Other Pre Specified Outcome: Anti-P. Gingivalis IgG in Serum
Description: Anti-P. gingivalis immunoglobulin G (IgG) in serum
  Antibody levels were measured by ELISA and outcome measure are ELISA UNITS (EU)
  Lower levels represent a pharmacodynamic effect of the drug on its target
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: EU
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 212 | 217
EU
  Baseline: number analyzed (Participants) | 213 | 209 | 212
  Baseline | 191.6 (216.8) | 202.4 (214.0) | 193.1 (199.5)
  Week 48: number analyzed (Participants) | 130 | 131 | 167
  Week 48 | 77.8 (123.2) | 110.8 (184.3) | 134.4 (201.0)

7. Other Pre Specified Outcome: Magnetic Resonance Imaging
Description: Change in magnetic resonance imaging - bilateral whole brain volume
  Larger volume may represent effect of the drug on its target
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: volume (CM^3)
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 214 | 212 | 217
volume (CM^3)
  Baseline: number analyzed (Participants) | 198 | 199 | 202
  Baseline | 1005154 (106682) | 1008135 (105765) | 1001711 (111145)
  Week 48: number analyzed (Participants) | 105 | 113 | 141
  Week 48 | 982782 (111888) | 987998 (102961) | 986119 (111779)

8. Other Pre Specified Outcome: Periodontal (or Gum) Pocket Depth
Description: Periodontal (or gum) pocket depth - pocket depth for only sites with depth >= 4mm.
  The primary endpoint was mean change in pocket depth from baseline to the end of the double-blind treatment period for tooth sites with depth ≥ 4mm at any time during the study. Therefore, values presented may be less than 4mm.
  Larger measure means worse outcome
Time Frame: Baseline to Week 48
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
Number analyzed (Participants) | 79 | 64 | 77
mm
  Baseline | 4.04 (0.75) | 4.03 (0.59) | 3.74 (0.66)
  Week 48: number analyzed (Participants) | 39 | 31 | 54
  Week 48 | 3.67 (0.92) | 3.78 (0.71) | 3.57 (0.61)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from screening through 48 weeks of treatment and 6 weeks of follow up, a total of approximately 60 weeks.
Arm/Group | COR388 80 mg BID (Twice Daily) | COR388 40 mg BID (Twice Daily) | Placebo BID (Twice Daily)
All-Cause Mortality (participants affected / at risk) | 5/214 | 1/212 | 0/217
Serious Adverse Events (participants affected / at risk) | 25/214 | 20/212 | 19/217
Other Adverse Events (participants affected / at risk) | 139/214 | 150/212 | 88/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COR388 80 mg BID (Twice Daily) (N=214) | COR388 40 mg BID (Twice Daily) (N=212) | Placebo BID (Twice Daily) (N=217)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
general physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0)
abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
multiple fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
liver function test abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
psychotic behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COR388 80 mg BID (Twice Daily) (N=214) | COR388 40 mg BID (Twice Daily) (N=212) | Placebo BID (Twice Daily) (N=217)
abdominal pain (Gastrointestinal disorders) | 11 | 7 | 3
diarrhea (Gastrointestinal disorders) | 27 | 34 | 7
nausea (Gastrointestinal disorders) | 13 | 13 | 4
decreased appetite (Metabolism and nutrition disorders) | 10 | 9 | 2
ALT increased (Investigations) | 37 | 20 | 4
AST increased (Investigations) | 34 | 20 | 3
amylase increased (Investigations) | 16 | 12 | 8
lipase increased (Infections and infestations) | 20 | 13 | 11
headache (Nervous system disorders) | 15 | 18 | 14
agitation (Psychiatric disorders) | 10 | 9 | 7
fall (Injury, poisoning and procedural complications) | 11 | 7 | 5
urinary tract infection (Infections and infestations) | 28 | 16 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators and/or their associates may publish findings of this study in scientific journals or present them at scientific meetings, provided the Sponsor is given ample opportunity to review any proposed abstract, manuscript, or slide presentation before its submission.

DOCUMENTS (2):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03823404/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03823404/SAP_001.pdf